CLINICAL TRIAL: NCT05186857
Title: Impact of Intestinal Metabolome and Microbiome Disbalance of Recipients of Hematopoietic Transplant in the Development of Acute Graft Versus Host Disease.
Brief Title: Metabolome and Microbiome Impact on Acute GVHD in Recipients of Hematopoietic Transplant
Acronym: AlloBolome
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: AlloBolome
Record Dates: First submitted 2021-11-29; First posted 2022-01-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Graft-versus-host Disease
Keywords: Acute graft-versus-host disease; Microbiome; Metabolome; Hematopoietic transplant
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent published data suggest that specific alterations in intestinal metabolome signature of hematopoietic stem cell transplant (allo-SCT) recipients might influence incidence and severity of acute graft versus host disease (aGVHD). Nevertheless, this possible relationship has not been undoubtedly established, pathophysiologic mechanisms have not been elucidated and possible clinical implications have not been studied. We hypothesized that in the early phase of allo-SCT, specific alterations in faecal metabolome occurred related to loss of intestinal microbiota diversity and disbalance of specific bacterial taxa, and that both alterations determine reduced survival of patients through increased incidence and severity of aGVHD. To test this hypothesis, a prospective multi-center cohort of allo-SCT recipients will had faecal and plasmatic samples collected at predetermined time-points pre&post-allo-SCT, and clinical relevant variables will be prospectively recorded throughout two years posttransplant follow-up. Metabolomic and microbiome analysis will be done to answer objectives of the study. To additionally explore if differential evolving characteristics in the intestinal metabolome and microbiome of donor/recipient sibling pairs influence the incidence and severity of aGVHD, probability of malignancy relapse and early and late mortality an additional cohort of family donors of enrolled patients will also have faecal and plasmatic samples collected and analysed.

ELIGIBILITY:
Patients Patients receiving an allotransplant at participating hospitals during the study period before initiating conditioning period.

Inclusion Criteria:

* Patients of any age who will receive allogeneic hematopoietic transplantation of any modality with any diagnosis.
* Agreement of the patient to participate by signing the informed consent or his/her legal representatives/assent (if applicable).

Exclusion Criteria

- Allotransplant recipients in stages after the initial pre-conditioning.

Donors

Family donors from patients included in the study:

Inclusion criteria:

* Agreement of the donor to participate by signing the informed consent or his/her legal representatives/assent (if applicable).
* Donor relatives with any degree of identity in the Human Leukocyte Antigens (HLA).

Exclusion Criteria:

* Unrelated donors
* Transplants from umbilical cord blood source.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving an allotransplant and family donors of the included patients.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Metabolome | From pre-Conditioning (Day -15) to Day +100 post-transplant.
  Sequential pre-transplant/post-transplant modifications in faecal and plasmatic levels of: 1.a. Butyrate (targeted analysis), 1.b: Biliary acids (targeted analysis) and 1.c. Metabolomic signature (untargeted analysis).
Incidence of Acute graft versus host disease | From the day of transplant (Day 0) to Day +100 posttransplant.
  Comparison of the incidence of any degree, degree-II and degree-III/IV of acute graft versus host disease between sub-groups of patients defined according to obtained metabolome results.
Overall Survival | From the day of transplant (Day 0) to 2 years posttransplant.
  Comparison of overall survival between obtained groups according to metabolome results.
Disease free survival | From the day of transplant (Day 0) to 2 years posttransplant.
  Comparison of overall survival between obtained groups according to metabolome results.

SECONDARY OUTCOMES:
Microbiome (alpha diversity of the intestinal microbiota) | At Day -15 and Day +30 post-transplant.
  Comparison of biological alpha diversity of the intestinal microbiota. Calculation of alpha diversity (Shannon's diversity index, observed OTUs, Faith's Phylogenetic Diversity and Evenness) index by QIIME-
Microbiome (beta diversity of the intestinal microbiota) | At Day -15 and Day +30 post-transplant.
  Comparison of biological beta diversity of the intestinal microbiota. Calculation of beta diversity (Jaccard distance, Bray-Curtis distance, Unweighted UniFrac distance and Unweighted UniFrac distance) index by QIIME-
Microbiome (alpha diversity of the plasmatic microbiota) | At Day -15 and Day +30 post-transplant.
  Comparison of biological alpha diversity of the plasmatic microbiota. Calculation of alpha diversity (Shannon's diversity index, observed OTUs, Faith's Phylogenetic Diversity and Evenness) index by QIIME-
Microbiome (beta diversity of the plasmatic microbiota) | At Day -15 and Day +30 post-transplant.
  Comparison of biological beta diversity of the plasmatic microbiota. Calculation of beta diversity (Jaccard distance, Bray-Curtis distance, Unweighted UniFrac distance and Unweighted UniFrac distance) index by QIIME-
Relapse | From the day of transplant (Day 0) to +30, +100, +365 and two years posttransplant.
  Comparison of patients´s incidence of relapse of the malignant disease between the groups obtained according to microbiome-metabolome results.
Mortality | From the day of transplant (Day 0) to Days +30, +100, +365 and two years posttransplant.
  Comparison of patients mortality between the groups obtained according to microbiome-metabolome results.

CONTACTS AND LOCATIONS:
Overall Officials: Ildefonso Espigado, PhD, Principal Investigator — Seville University, Dep. of Medicine. Virgen del Rocío/Virgen Macarena Hospitals, Instituto de Investigación Biomédica de Sevilla / CSIC, Seville, Spain
Locations (9):
- Spain (9):
  - Hospital Marqués de Valdecillas, Santander, Santander, Cantabria
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Virgen de las Nieves de Granada, Granada, Granada
  - Hospital del Niño Jesús, Madrid, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid, Madrid
  - Hospital Regional Universitario de Málaga, Málaga, Málaga
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Sevilla, Seville, Seville
  - Hospital Clínico de Valencia, Valencia, Valencia